CLINICAL TRIAL: NCT00201513
Title: Randomized Controlled Trial of Stabilizing Exercises and Effect on Anticipatory Muscle Control in Patients With Subacute and Chronic Low Back Pain
Brief Title: Anticipatory Muscle Control and Effect of Stabilizing Exercises in Patients With Subacute and Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Norwegian Fund for Postgraduate Training in Physiotherapy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REK 4.2005.1720
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Low Back Pain
Keywords: Muscle, Skeletal; Neuromuscular control; Stability; Exercise; Anticipatory muscle control
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TrA exercise (Experimental): Isolated Transversus abdominis (TrA) exercises (low load)
  Interventions: Behavioral: Isolated Transversus abdominis (TrA) exercise
- sling exercise (Experimental): Sling exercises (high load)
  Interventions: Behavioral: sling exercise
- group exercise (Active Comparator): Non-specific group exercises
  Interventions: Behavioral: group exercise

INTERVENTIONS:
Behavioral: Isolated Transversus abdominis (TrA) exercise — Eight weeks Isolated Transversus abdominis (TrA) exercise(low load) program; Isolated TrA control through biofeedback
  Arms: TrA exercise
Behavioral: sling exercise — Eight weeks sling(high load) exercise program; Isolated TrA control through biofeedback
  Arms: sling exercise
Behavioral: group exercise — Eight weeks non-specific group exercise program; Isolated TrA control through biofeedback
  Arms: group exercise

SUMMARY:
Muscular stability is essential to the spinal column to avoid harmful strain and injury to its structures. Sudden postural disturbances impose reactive internal forces through the spine. If the muscles do not react before the internal reactive forces propagate through the spine, there is a short fraction of time where the spinal column may lack sufficient muscular support. Studies have shown that in patients with low back pain deep abdominal and back muscle have a delayed response to reactive forces. The purpose of this study is to verify these findings and to investigate whether tailored interventions can improve the reaction time in stabilizing muscle around the lower spinal column i patients with subacute and chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Unspecific subacute, subacute remitting and chronic LBP
* Both sexes, 20-60 yrs of age
* LBP between 2-8 on a 11-pt numeric rating scale

Exclusion Criteria:

* Previous back surgery
* Sick listed more than one year
* Radiating pain below knee or motor deficits
* Systemic diseases and "red flags"
* Diagnosed psychiatric disease
* Ingoing insurance claim
* Pregnancy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2006-01; Primary Completion 2007-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Muscle activity onset in transversus abdominal muscle | 1 year

SECONDARY OUTCOMES:
Pain | 2 years
Function (Oswestry v2) | 2 years
Fear of avoidance belief | 1 year
Assessment of isolated transversus abd. and multifidus control | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ottar Vasseljen, PhD, Study Chair — National center for spinal diseases
Locations (1):
- Norwegian University of Science and Technology, National center for spinal diseases, Trondheim, Trondheim, Norway

REFERENCES:
- [Result] Unsgaard-Tondel M, Fladmark AM, Salvesen O, Vasseljen O. Motor control exercises, sling exercises, and general exercises for patients with chronic low back pain: a randomized controlled trial with 1-year follow-up. Phys Ther. 2010 Oct;90(10):1426-40. doi: 10.2522/ptj.20090421. Epub 2010 Jul 29. PMID 20671099
- [Result] Vasseljen O, Fladmark AM. Abdominal muscle contraction thickness and function after specific and general exercises: a randomized controlled trial in chronic low back pain patients. Man Ther. 2010 Oct;15(5):482-9. doi: 10.1016/j.math.2010.04.004. PMID 20621545
- [Result] Vasseljen O, Unsgaard-Tondel M, Westad C, Mork PJ. Effect of core stability exercises on feed-forward activation of deep abdominal muscles in chronic low back pain: a randomized controlled trial. Spine (Phila Pa 1976). 2012 Jun 1;37(13):1101-8. doi: 10.1097/BRS.0b013e318241377c. PMID 22146280
- [Derived] Unsgaard-Tondel M, Lund Nilsen TI, Magnussen J, Vasseljen O. Is activation of transversus abdominis and obliquus internus abdominis associated with long-term changes in chronic low back pain? A prospective study with 1-year follow-up. Br J Sports Med. 2012 Aug;46(10):729-34. doi: 10.1136/bjsm.2011.085506. Epub 2011 Jul 26. PMID 21791459